CLINICAL TRIAL: NCT02650791
Title: Platelet Transfusion Requirements in Hematopoietic Transplantation(PATH Pilot)
Brief Title: Platelet Transfusion Requirements in Hematopoietic Transplantation Pilot Study
Acronym: PATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20150629-01H
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic Platelet Transfusions (No Intervention): Patients allocated to the prophylactic platelet transfusion group will receive a platelet transfusion when the measured platelet count is less than 10 x 10^9/L.
- Prophylactic Tranexamic Acid (Experimental): Patients allocated to the prophylactic Tranexamic Acid group will receive a standardized routine oral dose of Tranexamic Acid 1 gram three times daily. Tranexamic Acid will start when Platelet count is less than 50 x 10^9/L and continue until platelet engraftment. Patients in this group will not receive routine prophylactic platelet transfusions
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Prophylactic Tranexamic Acid

SUMMARY:
It is hypothesized that a strategy using prophylactic oral Tranexamic Acid (TXA) with therapeutic platelet transfusions is safe and effective compared to prophylactic platelet transfusions in patients undergoing an autologous hematopoietic stem cell transplantation (who are at risk for bleeding).

DETAILED DESCRIPTION:
In Canada, over 1,500 autologous hematopoietic stem cell transplantations (ASCT) are performed annually for hematologic malignancies. It is currently standard practice to provide a prophylactic transfusion of platelets to prevent bleeding when the daily measured platelet count is less than 10 x 109/L. A patient may require up to six adult platelet doses during the post-transplant period. However, the true benefit of prophylactic platelet transfusions in the ASCT setting is unclear and has been called into question by several recent studies.

Prophylactic platelet transfusions may not only be unnecessary, they may be detrimental to the patient. Among blood products, platelet transfusions are associated with the highest risk of both infectious and non-infectious complications: this would include bacterial infections and allergic /febrile reactions. Moreover, the potential overuse of platelet products places a significant burden on a scarce health care resource that is provided through volunteer donations.

An alternative strategy to prevent bleeding and reduce the need for platelet transfusions involves administering Tranexamic Acid, an oral antifibrinolytic agent to stabilize blood clots and reduce bleeding. Tranexamic Acid is safe and effective in many clinical scenarios, and may be a reasonable alternative for prophylactic platelet transfusions. In the setting of ASCT, Tranexamic Acid may reduce bleeding and further enhance a strategy of therapeutic platelet transfusions where platelets are administered only in the event of active bleeding symptoms.

The effect of prophylactic platelet transfusions and Tranexamic Acid on clinical, quality of life and economic outcomes in patients receiving ASCT is unknown. The primary aim of this research program is to perform a randomized controlled trial to determine whether a strategy of prophylactic Tranexamic Acid (with therapeutic platelet transfusions) is safe and effective compared to prophylactic platelet transfusions in patients undergoing ASCT. Before conducting a larger trial, the investigators first propose a pilot randomized controlled trial to determine the feasibility of such a study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are aged 18 years old or older and undergoing an autologous HSCT (hematopoietic stem cell transplantation) for any hematologic malignancy.

Exclusion Criteria:

1. A previous WHO grade 3 or 4 bleeding event
2. A WHO grade 2 bleeding event within the past year
3. A previous or current unprovoked thrombotic event defined as a pulmonary embolism, deep vein thrombosis, cerebral thrombosis
4. Current or previous (within 2 weeks) urinary tract bleeding
5. An inherited hemostatic or thrombotic disorder
6. Coagulopathy defined as a prothrombin time or activated partial thromboplastin time >1.5 times the upper limit of normal or fibrinogen less than 2 g/L
7. A requirement for therapeutic anticoagulant or antiplatelet drugs
8. Previously documented history of refractoriness to platelet transfusion secondary to HLA (Human Leukocyte Antigen) antibodies
9. Significant renal impairment (creatinine >1.5 times the upper limit of normal)
10. Pregnant or breast-feeding
11. Unwilling or unable to provide informed consent
12. Participant has ever had a pulmonary embolism, deep vein thrombosis, cerebral thrombosis or has active angina
13. Participant has known history of subarachnoid hemorrhage
14. Participant has acquired disturbances to his/her colour vision
15. Participant has known sensitivity or allergy to Tranexamic Acid or any of its ingredients
16. The current use of oral contraceptive pill (Birth Control Pill), hormonal contraceptives or hormone replacement therapy .

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Enrolment, as measured by the number of patients screened per month at each site | monthly, up to 23 months
Number of off-protocol platelet transfusions, with a target of < 10% off-protocol transfusions in each treatment arm | monthly, up to 23 months
Total number of platelet transfusions/group, with a target of 25% reduction in the tranexamic acid arm | monthly, up to 23 months
Adherence to tranexamic acid use, defined as excellent (greater than or equal to 90% use), acceptable (75-90% use), poor (< 75% use) | monthly, up to 23 months

SECONDARY OUTCOMES:
WHO (World Health Organization) Bleeding events of Grade 2 or higher | daily, up to one month
Time from randomization to bleeding of WHO bleeding events Grade 2 or higher | daily, up to one month
Number of days with bleeding of WHO bleeding events Grade 2 or higher | daily, up to one month
Bleeding Severity Measurement Scale for bleeding events Grade 2 or higher | daily, up to one month
Number of platelet and/or red cell transfusions | daily, up to one month
Time to platelet recovery | daily, up to one month
Number of days with platelet count < 10 x 10^9/L | daily, up to one month
LOS (Length of hospital stay) | Length of stay will be measured as the number of days elapsed between hospital admission and hospital discharge dates up to 1 month
  LOS=discharge date - admission date
Adverse transfusion reactions | daily, up to one month
  Number and type of reactions will be recorded.
Bearman Toxicity Score | Day 30
  Validated scoring system to assess toxicity during stem cell transplantation
Infections at Day 30 | Day 30
Quality of Life measurements, as determined by a battery of QoL instruments | daily, up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tinmouth, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Hamilton Health Sciences - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tay J, Allan D, Beattie S, Bredeson C, Fergusson D, Maze D, Sabloff M, Thavorn K, Tinmouth A. Rationale and design of platelet transfusions in haematopoietic stem cell transplantation: the PATH pilot study. BMJ Open. 2016 Oct 24;6(10):e013483. doi: 10.1136/bmjopen-2016-013483. PMID 27798034